CLINICAL TRIAL: NCT04013048
Title: A Phase I Mass Balance and Biotransformation Study of [14C]-Fluzoparib in Chinese Patients With Solid Tumor
Brief Title: Study to Evaluate the Mass Balance and Biotransformation of [14C]-Fluzoparib in Chinese Patients With Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FZPL-I-107
Record Dates: First submitted 2019-07-07; First posted 2019-07-09 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2019-07

CONDITIONS: Solid Tumor
Keywords: Solid Tumor; 14C-Fluzoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]-Fluzoparib (Experimental): Patients will receive single dose of [14C]- Fluzoparib.
  Interventions: Drug: [14C]-Fluzoparib

INTERVENTIONS:
Drug: [14C]-Fluzoparib — Patients will receive single dose of orally [14C]- Fluzoparib on Day 1.

SUMMARY:
Study to Evaluate the Mass Balance and Biotransformation of Single Dose [14C]-FZPL in Chinese Patients with Solid Tumor

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed with advanced solid malignancies who are refractory or intolerant to standard therapy or considered to be benefit from the treatment of fluzoparib.
2. ECOG performance status of 0 to 1.
3. Life expectancy of more than 3 months.
4. Signing the informed consent forms.
5. Adequate bone marrow, liver and renal function.
6. Be able to communicate well with the researcher and be able to complete the trial in accordance with the program.

Exclusion Criteria:

1. Subjects who take any drugs that strongly inhibit or induce the CYP450 enzyme 14 days prior to study drug administration；
2. Those who have history of alcohol abuse (it was defined as that the daily alcohol consumption was higher than the following criteria: the weekly alcohol consumption was higher than 14 units of alcohol (1 unit= 360 ml beers/45 ml liquor containing 40% alcohol/150ml grape wine) 6 months prior to screening period, or the alcohol breath test results ≥20 mg/dl during screening period；
3. Subjects who smoked daily >5 sticks of cigarette 3 months prior to first dose or cannot give up smoking during study.
4. Subjects who have history of drug abuse or taking soft drug (i.e., marihuana) 3 months prior to screening period or taking hard drugs (i.e., cocaine, amphetamines, benzodiazepine, etc.); or the results of urine test in drugs were positive.
5. Subjects who were used to drink grapefruit juice or overconsumption of tea, coffee, and the drink with caffeine; and cannot give up them during test.
6. Subjects who need long-term exposure to radiation, or who have been exposed to PET-CT or ECT within 3 months prior to study drug administration or who have participated in the labeling test of radiopharmaceuticals.
7. Subjects who have fertility planning within the range of starting trial - 1 year after finishing trial.
8. Subjects who have excessive bleeding or blood donation (400ml) 3 months prior to screening period, or planned to donate blood 1 month after finishing this trial.
9. Subjects who have habitual constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease.
10. Subjects must not have had prior treatment with PARP inhibitors.
11. Subjects who cannot complete this study because of other reasons, or any factors judged by investigator that the participants cannot meet.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2019-12-24 (Actual)

PRIMARY OUTCOMES:
The distribution of Fluzoparib in the whole blood and plasma and whole.radioactive pharmacokinetics following the single orally administered [14C]-Fluzoparib in Chinese patients with advanced solid tumor. | Up to 10 days (approx) from the start of administration.
  The percentage of radioactive dose of [14C] radiolabelled Fluzoparib recovered in blood and in total, up to Day 10 (approx).
Quantitive analysis of whole radioactivity of excrement of orally administered [14C]-Fluzoparib in Chinese patients with advanced solid tumor to obtain the mass balance data and the main excretion pathway in human body. | Up to 10 days (approx) from the start of administration.
  The percentage of radioactive dose of [14C] radiolabelled Fluzoparib recovered in urine, faeces and in total, up to Day 10 (approx).
Identification of the main metabolite and biotransformation pathway of Fluzoparib and investigation of metabolite with proportion >10% in plasma following the single orally administered [14C]-Fluzoparib in Chinese patients with advanced solid tumor. | Up to 10 days (approx) from the start of administration.
  Proportion of different metabolites.
Quantitive analysis of the concentrations of Fluzoparib in plasma using the validated LC-MS/MS to obtain pharmacokinetic data. | Up to 10 days (approx) from the start of administration.
  The concentrations of Fluzoparib in plasma up to Day 10.
Observation of safety following the single orally administered [14C]-Fluzoparib in Chinese patients with advanced solid tumor. | Up to 10 days (approx) from the start of administration.
  Adverse events assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided